CLINICAL TRIAL: NCT02826642
Title: A Phase I, Open Label, Multicenter, Dose Finding Study of IDH305 With Standard of Care in IDH1 Mutant Acute Myeloid Leukemia
Brief Title: A Dose Finding Study of IDH305 With Standard of Care in IDH1 Mutant Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIDH305X2102
Record Dates: First submitted 2016-06-13; First posted 2016-07-11 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: newly diagnosed acute myeloid leukemia; AML; myeloid dysplastic syndrome; MDS; IDH305; standard of care in IDH1 mutant acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Medically fit for induction (Experimental): IDH305 + Standard of care for patients that are medically fit for induction.
  Interventions: Drug: IDH305
- Arm 2 Medically unfit for induction (Experimental): IDH305 + Standard of care for patients that are medically unfit for induction.
  Interventions: Drug: IDH305

INTERVENTIONS:
Drug: IDH305

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and potential efficacy of IDH305 with standard treatments for newly diagnosed IDH1R132 mutant acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

-- Previously untreated AML. Patients with untreated, high or very high risk MDS (according to rIPSS or equivalent) are also permitted in Arm 2.

* Documentation of IDH1R132 mutation of tumor
* ECOG performance status ≤ 2
* Clinically fit for standard of care medication per protocol.

Exclusion Criteria:

* Prior treatment for AML or MDS
* Any severe or uncontrolled medical conditions that would prevent the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures such as the presence of other clinically significant cardiac, respiratory, gastrointestinal, renal, hepatic or neurological disease.
* Acute Promyelocytic Leukemia
* Women who are pregnant or lactating

Other protocol-defined Inclusion/Exclusion may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2016-11-29 (Estimated); Study Completion 2016-11-29 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting toxicities | 10 months
  (escalation only)
Number of patients with adverse events (AEs) | 36 months

SECONDARY OUTCOMES:
Area Under Curve (AUC) | 36 months
  To characterize the PK profile of IDH305 with SOC medications (each Arm)
Maximum Plasma Concentration (Cmax) | 36 months
  To characterize the PK profile of IDH305 with SOC medications (each Arm)
Time taken to reach maximum plasma concentration (Tmax) | 36 months
  To characterize the PK profile of IDH305 with SOC medications (each Arm)
Complete remission rate (CRR) | 36 months
  To characterize preliminary anti-tumor activity for each arm of the study. (Arm 1 and Arm 2)
Overall response rate (ORR) | 36 months
  To characterize preliminary anti-tumor activity for each arm of the study. (Arm 1 and Arm 2)
Event free survival (EFS) | 36 months
  To characterize preliminary anti-tumor activity for each arm of the study. (Arm 1 and Arm 2)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals